CLINICAL TRIAL: NCT03664336
Title: Refractory Diffuse Large B-cell Lymphoma After First-line Immuno-CT: Treatment Options and Outcomes
Brief Title: Refractory Diffuse Large B-cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: refractory DLBCL
Record Dates: First submitted 2018-08-22; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: diffuse large B-cell lymphoma; refractory; rituximab
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the rituximab era, one-third of diffuse large B-cell lymphoma (DLBCL) patients experience relapse/refractory disease after first-line anthracycline-based immunochemotherapy (IChemo). Optimal management remains an unmet medical need. The aim of this study was to report the outcomes of a cohort of refractory patients according to their patterns of refractoriness and the type of salvage option. The investigators performed a retrospective analysis, which included 104 DLBCL patients treated at Lyon Sud University Hospital (2002-2017) who presented with refractory disease. The investigators retrospectively evaluated the outcomes of a cohort of 104 refractory patients according to their patterns of refractoriness and the type of salvage option.

ELIGIBILITY:
Inclusion Criteria:

-≥18 years of age

* diagnosed with DLBCL at Lyon Sud University Hospital (LSUH) from January 2002 to January 2017
* presented with refractory disease in response to front-line therapies
* including anthracycline-based chemo and a monoclonal anti-CD20 antibody

Exclusion Criteria:

* Patients with a history of indolent lymphoma,
* Patients with a primary central nervous system (CNS) lymphoma or immunosuppression-related lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Man or woman diagnosed for a DLBCL from January 2002 to January 2017
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Outcome according to pattern of refractoriness | Up to 4 years
  OS was defined as the time from first relapse, or progression, to death from any cause.

SECONDARY OUTCOMES:
Outcome according to pattern of refractoriness | Up tp 24 months
  EFS was defined as the time from first relapse, or progression, to the next event (defined as either second relapse/progression, change of therapy, or death from any cause). Patients who did not experience an event were censored at the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Clémentine Sarkozy, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France